CLINICAL TRIAL: NCT00347412
Title: Phase 3 Trial, Randomized, Open-Label, of NOV-002 in Combination With Paclitaxel and Carboplatin vs. Paclitaxel and Carboplatin Alone for the Treatment of Advanced Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Study of NOV-002 in Combination With Chemotherapy to Treat Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NOV002-C301
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Stage IIIb; Stage IV; Non Small Cell Lung Cancer (NSCLC); NSCLC Stage IIIb with malignant pleural/pericardial effusion; NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pericardial Effusion | interventions — Paclitaxel; Albumin-Bound Paclitaxel; NOV 002; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: NOV-002 plus Chemotherapy (Experimental): NOV-002 in combination with Paclitaxel and Carboplatin
  Interventions: Drug: Paclitaxel; Drug: NOV-002; Drug: Carboplatin
- Group B: Chemotherapy Alone (Active Comparator): Paclitaxel and Carboplatin
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel is dosed at 200 mg/m2, as a 3 hour infusion.
  All randomized patients will follow the established 21-day cycle of paclitaxel and carboplatin including the administration of pre-medications for these products per the package inserts. Paclitaxel and carboplatin cycles will be administered until documented disease progression or completion of 6 cycles of paclitaxel and carboplatin in the absence of response or unacceptable related toxicity, whichever comes first.
  Other Names: Abraxane; Onxol; Taxol
Drug: NOV-002 — * Two 60 mg intravenous boli given 3 hours apart administered the day prior to the first administration of paclitaxel and carboplatin cycle one
  * For each nominal 21-day paclitaxel and carboplatin cycle:
    * 60 mg given intravenously on Day 1, given one hour prior to paclitaxel and carboplatin
    * followed by 60 mg subcutaneously daily for the next 20 days. If there is a delay in chemotherapy cycles, the patient will continue with daily, subcutaneous administration of NOV-002 until the next cycle of chemotherapy begins
  Patients randomized to NOV-002 Group A, will receive NOV-002 until disease progression, unacceptable NOV-002 related toxicity, or discontinuation of paclitaxel and carboplatin, whichever comes first.
  Arms: Group A: NOV-002 plus Chemotherapy
Drug: Carboplatin — Carboplatin is dosed at an area under the curve (AUC) of 6 mg/mL/min using the Calvert equation for carboplatin dosing.
  All randomized patients will follow the established 21-day cycle of paclitaxel and carboplatin including the administration of pre-medications for these products per the package inserts. Paclitaxel and carboplatin cycles will be administered until documented disease progression or completion of 6 cycles of paclitaxel and carboplatin in the absence of response or unacceptable related toxicity, whichever comes first.
  The initial dose of chemotherapy for every patient in the trial is 200 mg/m2 of paclitaxel, as a 3 hour infusion, followed by carboplatin at an area under the curve (AUC) of 6 mg/mL/min using the Calvert equation for carboplatin dosing.
  Other Names: Paraplatin

SUMMARY:
The purpose of this clinical trial is to find out whether or not the combination of NOV-002 with chemotherapy (paclitaxel and carboplatin) is better at improving overall survival time when compared to chemotherapy alone in people with non-small cell lung cancer (NSCLC).

Earlier clinical trials in NSCLC showed that patients treated with NOV-002 in combination with chemotherapy had a better response (their tumors got smaller in one United States Phase 1/2 trial) than patients who received chemotherapy alone; and in two Phase 2 trials done in Russian patients, at the end of one year, patients treated with NOV-002 with chemotherapy had a better survival rate than patients who did not receive NOV-002 with their chemotherapy.

DETAILED DESCRIPTION:
NSCLC is a widespread disease with extremely high mortality and morbidity. Even the most widely accepted standard of care chemotherapy in advanced NSCLC, platinum-based doublets, are only palliative, providing marginal efficacy as measured by survival. In addition, such chemotherapy is accompanied by severe, sometimes life-threatening, toxicities which often limit its application. Thus, there is a clear need for new, more effective and safer therapies for advanced NSCLC. In Phase 2 trials, NOV-002 demonstrated a higher response rate and improved survival compared to chemotherapy alone in patients with advanced NSCLC, and was well-tolerated in this patient group. Thus, we are conducting a large Phase 3 trial of NOV-002 to better define its clinical profile and potential benefit in advanced NSCLC patients.

The overall design of this Phase 3 trial reflects major elements of the previous Russian and US clinical trials in advanced NSCLC - it is an open label, randomized controlled trial comparing NOV-002 in combination with first-line chemotherapy (paclitaxel + carboplatin) to first-line chemotherapy alone. Furthermore, it is designed and powered to be a pivotal, registrational trial, sufficient for approval. As its primary efficacy endpoint, this Phase 3 trial aims to demonstrate that the combination of NOV-002 with paclitaxel and carboplatin results in improved overall survival when compared with paclitaxel and carboplatin alone. In addition, several secondary efficacy endpoints will be assessed, including progression free survival, tumor response rate and duration of response, quality of life, myelosuppression and immunomodulation. Overall survival was chosen as the primary endpoint of this trial in the context of FDA (Draft) Guidance ("Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics", April 2005). This Guidance indicates that an improvement in overall survival should be evaluated in randomized controlled trials and is of unquestioned clinical benefit. It indicates that the endpoint is precise and easy to measure, documented by the date of death, and states that bias is not a factor in endpoint measurement, and blinding is not essential. This Phase 3 randomized, controlled, open-label trial thus conforms to this Guidance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage IIIb with malignant pleural or pericardial effusion or Stage IV (American Joint Committee on Cancer [AJCC]) NSCLC
* ECOG performance score of 0 or 1
* Adequate bone marrow, hepatic, and renal function
* New York Heart Association (NYHA) score 1-2
* Life expectancy of at least 12 weeks
* Women of child-bearing potential and men whose partners are of child-bearing potential must be willing to use an acceptable method of birth control during trial participation or are surgically sterile or women who are post-menopausal (defined as not having a menstrual cycle for greater than two years).
* The patient or patient's legal representative has the ability to understand the requirements of the trial, has provided written informed consent, and agrees to abide by the trial restrictions and to return for the required assessments.
* The patient must be able to self administer daily subcutaneous injections or his/her caregiver must be able to administer daily subcutaneous injections.

Exclusion Criteria:

* Prior chemotherapy for advanced NSCLC or the patient has received prior neoadjuvant or adjuvant chemotherapy for NSCLC in the year prior to the date of randomization
* Patients with central nervous system (CNS) metastases
* Any systemic disease precluding chemotherapy
* Chronic use of systemic corticosteroids in pharmacological doses
* Known or history of HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Contraindication to treatment with paclitaxel or carboplatin or any of the components of NOV-002
* Any known preexisting medical condition, including substance abuse, that could interfere with the patient's participation in and completion of the protocol
* Have received any investigational drug, defined as a drug for which there is no Food and Drug Administration (FDA) approved indication, within the 30 days prior to randomization
* Pregnant female or nursing mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Overall survival during the length of the trial, length of the trial is approximately two years after last patient in | 16 months

SECONDARY OUTCOMES:
Improved progression-free survival (PFS) | 16 months
Higher anti-tumor overall response rate (ORR) | 16 months
Less myelosuppression and improved recovery from chemotherapy-induced myelosuppression | 16 months
Immunomodulation as evidenced by changes in lymphocyte subsets | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lynch, MD, Study Chair — Massachusetts General Hospital; Panos Fidias, MD, Study Chair — Massachusetts General Hospital
Locations (75):
- United States (12):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Sharp Memorial Hospital, San Diego, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - St. Agnes Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Park Nicollet Clinic - Cancer Center St. Louis Park, Saint Louis Park, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cleveland Clinic Foundation Taussig Cancer Center, Cleveland, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - South Texas Institute of Cancer, Corpus Christi, Texas
- Canada (4):
  - William Osler Health Center, Brampton, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Laval Hospital, Sainte-Foy, Quebec
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Lin Clinic, Haifa
  - Meir Medical Center, Kfar Saba
  - Institute of Oncology, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Assaf Harofeh Hospital, Ẕerifin
- Italy (3):
  - Azienda Ospedaliera Treviglio Caravaggio, Bergamo
  - Azienda Ospedaliera Careggi, Florence
  - Sondrio Hospital, Sondrio
- Poland (10):
  - Oddzial Pulmonologiczny z Pododdzialem Chemioterapii, Bystra
  - Samodzielny Publiczny Szpital Kliniczny N°.1, Gdansk
  - Oddzial Chemioterapii Pomorskie Centrum Onkologii,, Gdynia
  - Katedra Onkologii Akademii Medycznej w Lodzi, Lodz
  - Oddzial Chemioterapii Zaklad Opieki Zdrowotnej MSWiA, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy Oddzial III, Otwock
  - Wielkopolskie Centrum Chorob, Poznan
  - Oddzial Gruzlicy I Chorob Pluc I P, Prabuty
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie w Warszawie, Warsaw
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
- Romania (5):
  - S.C. Oncomed SRL, Timișoara, Timiș County
  - Institute of Oncology, Department of Medical Oncology II, Bucharest
  - Institute of Oncology Cluj-Napoca, Cluj-Napoca
  - Institute of Oncology, Cluj-Napoca, Cluj-Napoca
  - Craiova Emergency Clinical County Hospital, Craiova
- Russia (15):
  - Arkhangelsk Regional Clinical Oncology Center, Arkhangelsk
  - Chelyabinsk Regional Oncology Center, Chemotherapy Department, Chelyabinsk
  - Clinical Oncology Center, Chemotherapy Department, Kazan'
  - Omsk Regional Clinical Oncology Center, Omsk
  - Orenburg Regional Clinical Oncology Center, Orenburg
  - Stavropol Regional Clinical Oncology Center, Pyatigorsk
  - Leningrad Regional Clinical Hospital, Department of Thoracic Surgery, Saint Petersburg
  - City General Hospital #2, City Center of Intensive Pulmonology and Thoracic Surgery, Saint Petersburg
  - St. Petersburg Pavlov State Medical University under the Federal Agency for Healthcare and Social Development, Saint Petersburg
  - City Clinical Oncology Center, Thoracic Department, Saint Petersburg
  - Oncology Center, Hematology Department, Sochi
  - Stavropol Regional Clinical Oncology Center, Chemotherapy Department, Stavropol
  - Tambov Regional Oncology Center, Chemotherapy Department, Tambov
  - Kazan Oncology Center, Tatarstan
  - Voronezh Regional Clinical Oncology Center, Voronezh
- Serbia (3):
  - Clinical Hospital Center Bezanijska kosa, Belgrade
  - Institute of Lung Diseases Sremka Kamenica, Kamenitz
  - Clinical Center Nis, Clinic for Lung Diseases "Knez Selo", Niš
- Spain (2):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Mutua de Terrassa, Terrassa
- Kantonales Spital Sursee-Wolhusen, Sursee, Switzerland
- Ukraine (8):
  - Cherkasy Regional Oncology Center, Cherkassy
  - Public Treatment and Prophylaxis Institution: Chernihiv Regional Oncology Center, Chernihiv
  - City General Hospital #4, Dnipropetrovsk
  - Regional Oncological Center, Ivano-Frankivsk
  - S.P. Grigoryev Institute of Medical Radiology, Kharkiv
  - Oncology Institute under the Ukrainian Academy of Medical Sciences, Kyiv
  - Crimean Republican Clinical Oncology Center, Simferopol
  - Zakarpatsky Regional Oncological Clinical Center, Uzhhorod
- United Kingdom (6):
  - Anchor Unit, Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital and Medical School Department of Cancer Medicine, Dundee, Scotland
  - St. Luke's Cancer Centre, Guildford, Surrey
  - Oncology Research, Nottingham City Hospital, Nottingham
  - Dorset Cancer Centre, Poole Hospital, Poole
  - Yeovil District Hospital NHS Foundation Trust, Higher Kingston, Somerset